CLINICAL TRIAL: NCT02061163
Title: Evaluation of Contrast-Enhanced Ultrasound in Human Crohn's Disease
Brief Title: Contrast-Enhanced Ultrasound in Human Crohn's Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI leaving UM at the end of the month
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jonathan R. Dillman M.D., Assistant Professor of Radiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00080030
Record Dates: First submitted 2014-02-06; First posted 2014-02-12 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — FS 069

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subjects with Crohn's disease (Experimental): Contrast Enhanced Ultrasound Optison
  Interventions: Device: Contrast Enhanced Ultrasound; Drug: Optison

INTERVENTIONS:
Device: Contrast Enhanced Ultrasound — Subjects with Crohn's disease will undergo contrast enhanced ultrasound imaging with shear wave elastography. Both CEUS and shear wave elastography will be performed using FDA approved ultrasound machines.
Drug: Optison — Optison is a microbubble contrast agent (dye) that will be injected during the CEUS imaging. Optison is FDA-approved for use in heart ultrasounds but not approved for use in bowel ultrasounds. Its use in this study is considered investigational (off-label).

SUMMARY:
To determine if contrast enhanced ultrasound (CEUS) and shear wave elastography can accurately diagnose bowel wall inflammation and fibrosis in patients with known Crohn's disease.

DETAILED DESCRIPTION:
Crohn's disease (CD) is an inflammatory condition that affects the intestinal tract (large and small bowels). Some patients with CD may get swelling of the intestinal tract (inflammation) or scarring of the intestinal tract (fibrosis). Fibrosis develops because of chronic injury. Both inflammation (swelling) and fibrosis (scarring) can cause the bowel to narrow, which can lead to the bowel becoming blocked. The long-term goal of this project is to develop new noninvasive radiology imaging tests that can show the difference between bowel wall inflammation and fibrosis. Currently there are no imaging tests that can do this reliably.

Current imaging methods (CT and MRI) that are ordered to help diagnose and follow-up CD are excellent at showing inflammation, but are not accurate for finding fibrosis. CT also exposes patients to small amounts of radiation, and both CT and MRI are costly. We are therefore studying ultrasound imaging, as it is more cost-effective and does not expose patients to radiation. CEUS uses microbubbles in a solution that are injected into a vein in one of the arms. This allows doctors to see the blood flow to parts of the body. This microbubble contrast agent (dye) is called Optison. Another imaging method, called shear wave elastography, uses sound waves to noninvasively measure the stiffness of structures in the body.

It is important to be able to tell the difference between inflammation and fibrosis in Crohn's disease, because narrowing of the bowel due to inflammation generally responds well to medications, whereas narrowing caused by fibrosis does not respond well to medications and may require surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 10 years of age and older
* Have been diagnosed with small bowel Crohn's disease
* Are receiving medical therapy for Crohn's disease
* Are scheduled for surgery (bowel resection) OR
* Are scheduled for a clinically-indicated MR enterography (MRE)/MRI exam.

Exclusion Criteria:

* Patients under the age of 10
* Are pregnant or breast feeding
* Are significantly overweight - BMI >35-40
* Have an inability to understand the consent
* Have prior allergic-like reaction or other adverse reaction to microbubble contrast agent
* Hypersensitivity to perflutren, blood, blood products or albumen
* Have a cardiac shunt
* Known unstable cardiac condition such as history of a heart attach, irregular heartbeat, congestive heart failure, etc.
* Known acute or chronic kidney disease, moderate/severe lung disease or acute or chronic liver disease

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of bowel wall inflammation and fibrosis in patients with Crohn's disease using CEUS | 2 years
  CEUS will be performed to evaluate inflammation and fibrosis in patients with Crohn's disease

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan C.S. Mott Children's Hospital, Ann Arbor, Michigan, United States